CLINICAL TRIAL: NCT04438161
Title: Identification of Newborns at High Risk for the Occurrence of Preventable Child Maltreatment: Phase 3 of Project 3 in the Overall Center for Innovation in Child Maltreatment Policy, Research, and Training (CICM), a Capstone Centers Grant.
Brief Title: Study to Understand Risk and Resilience Opportunity for Newborns After Delivery
Acronym: SURROuND
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Mini Tandon, Professor of Child and Adolescent Psychiatry, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202007199; 1P50HD096719 (NIH)
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: A. Longitudinal Cohort n=400; B. Lower Risk (n=45) and Higher Risk (n=105) Randomized 2:1 to PERCCS Intervention
Keywords: Child maltreatment, preventative intervention, case management, newborn, infancy
MeSH Terms: interventions — Community Support

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (study personnel blind to intervention allocation status)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Risk (Active Comparator): Low risk natural history study (n=250*)
  *Participants will be randomized 2:1 PERCCS:Control, and the randomization will be within successive sets of three families who fall in either "high risk" counts (n=105) families for child maltreatment or "low risk" counts (n=45) families.
  Interventions: Behavioral: PERCCS: Personalized Education Regarding Clinical and Community Supports
- High Risk (Experimental): High risk families in prospective longitudinal study of newborns (n=150*).
  *Participants will be randomized 2:1 PERCCS:Control, and the randomization will be within successive sets of three families who fall in either "high risk" counts (n=105) families for child maltreatment or "low risk" counts (n=45) families.
  Participants in this arm will be randomized to:
  1. PERCCS (see attached figure and table for details)
  2. Care as Usual
  Interventions: Behavioral: PERCCS: Personalized Education Regarding Clinical and Community Supports

INTERVENTIONS:
Behavioral: PERCCS: Personalized Education Regarding Clinical and Community Supports — A brief follow-up to the screening provided to 50% of the consented families (randomly assigned) that links their specific familial risks to community interventions.
  Other Names: Clinical and Community Supports

SUMMARY:
Childhood Maltreatment (CM) has highly deleterious effects on human development and is a preventable known cause of enduring psychopathology in the United States. Infants and young children are at particularly high risk for physical harm from abuse and neglect, comprising over 60% of all child maltreatment fatalities. An increasing number of studies point to the ability to target prevention of CM by estimating individual specific risk at the time of birth, on the basis of readily-accessible data elements of birth records. This clinical trial is a randomized controlled trial embedded within a prospective longitudinal study, in which families of infants recruited prenatally or in the newborn period are randomized to an enhanced level of engagement in resource navigation, which we refer to as Personalized Education Regarding Clinical and Community Supports (PERCCS). The enhancement involves keying recommendations for evidence-informed interventions for the prevention of CM to established risk factors for ascertained within a family.

The parent longitudinal cohort study involves enrollment of a diverse population of families of newborns (prenatally or in the immediate postnatal period) for the purpose of ascertaining sociodemographic, psychological (eg. parental stress) and family psychiatric risk factors for (a) child maltreatment (b) unmet service needs, and (c) adverse behavioral outcomes of the children. Families are contacted quarterly to track acquisition of support services that are relevant to the prevention of child maltreatment. At age 18 months early childhood behavioral outcomes are ascertained, biomaterials collected, and official-report child maltreatment records from the State of Missouri are individually cross-matched with identifiers of the children and their parents.

Two major outcomes are examined:

The first is whether the engagement protocol results in a higher level of acquisition and active participation in recommended preventive intervention services by the families (including home visitation, parental mental health care, evidence-based parenting education, and others delineated in Table 1, see below).

The second is the rate of child maltreatment (CM) ascertained in official Missouri state administrative records for which individual informed consent to individually-cross reference is obtained by the families in the course of their enrollment in the parent longitudinal study.

DETAILED DESCRIPTION:
Sample: The sample will be recruited from the Washington University School of Medicine Obstetrical Service within the Barnes Jewish Christian (BJC) Health System, on which there are over 3000 Missouri childbirths per year, serving an urban population of families that are disproportionately affected by poverty. Fifty-five per cent of patients report a family income less than $20,000, 65% of the mothers are unemployed, and the majority of the newborns are on Medicaid or are Medicaid-eligible. In preliminary screening efforts, over one third of the mothers reported their own childhood histories of maltreatment, and approximately one half score in the clinical range for depressive symptomatology.

Methods: A schematic summarizing study enrollment, participant randomization, and ascertainment of outcomes is provided in Figure 1.

Study Approach and Design: N=400 families are in the process of being enrolled in the parent longitudinal study. Among those who fall in an elevated risk category (upper 50% of the sample for total count of established risk factors) we will randomize 150 families 2:1 to Personalized Education Regarding Clinical and Community Supports (PERCCS) versus Usual Care. Risk counts are calculated by the total number of established predictors of risk for CM (itemized in Table 1) ascertained from birth records and: i) a screen for maternal depression, ii) a screen for maternal childhood trauma, and iii) a screen for active intimate partner violence. Utilization of community-based evidence-informed support services will be ascertained at baseline and quarterly thereafter for all study participants. Official-report Child Maltreatment data from Missouri state administrative data will be individually linked with participant research records when the children reach 18 months of age.

PERCCS involves i) a review with the mother of all family CM risks ascertained in the context of their own individual screening ii) recommendations of community and clinical interventions which substantively respond to those risks and are available to the subject (on the basis of each individual subject's zip code, insurance, and eligibility for the interventions), collectively the personalized family resource plan, iii) facilitation of contact between the subject and the respective provider agencies to initiate enrollment; and iv) authorization for the research team to share the personalized risk profile and support recommendations with the infant's outpatient primary care provider.

The community and clinical supports responsive to specific risk factors are listed in Table 1, which summarizes the array of evidence-informed preventions that will be presented to the families, and the correspondence with each to specific CM risks ascertained within a family. Table 2 depicts the set of scripts which are used by the study team to standardize all aspects of the review of endorsed risks, their potential adverse effects on parenting, and the opportunities for mitigation through evidence-informed intervention.

All participants will receive care as usual, including the provision of a summary document itemizing key community supports for families of infants, a continuously-updated local community resource handbook, a published parenting guide, and opportunity to enroll free-of-charge in a virtual parenting education and developmental surveillance program, babynavigator.com.

Key Measures:

The Utilization of Community Services (UCS) is a survey that will be used to ascertain engagement of families in community supports and interventions, including tracking of both frequency and duration. This survey is completed at the time of study enrollment to establish a baseline, and quarterly thereafter until the completion of the study when a child reaches 18 months of age.

State Records: The second primary outcome, rate of child maltreatment, will rely on official state records from the State of Missouri Department of Social Services. Participants are aware that accessing service records or CM report data are retrospective when acquired and do not pose any risk or liability to them nor can it impact services received.

Statistical Analyses:

I. Intent-to-treat analysis of impact of PERCCS on service utilization. We will calculate the total proportion of evidence-informed services indicated by risk profiles of all families within each group (the intervention group and the control group) and compare the groups using chi square analysis.

II. Intent-to-treat analysis of the impact of PERCCS on the occurrence of child maltreatment. We will compare the rate of official-report abuse/neglect between the groups using chi square analysis.

III. (Secondary) We will conduct logistic regression analysis simultaneously examining the effects of risk count and service access on official report child maltreatment outcome.

The randomized controlled trial has adequate statistical power to detect an odds ratio of 2.0 for the effect of PERRCS in reducing child maltreatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be Missouri residents
* 18 years of age or older
* Engaged in the BJC Healthcare Obstetrics or Newborn Services

Exclusion Criteria:

* Participants who are not Missouri residents
* Under the age of 18 years
* Not engaged in the BJC Healthcare Obstetrics or Newborn Services.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Service Utilization | Not more than 18 months postpartum
  Proportion of evidence-informed services indicated by risk profiles of all families within group acquired over the course of follow-up.
Child Maltreatment | Not more than 18 months postpartum
  Rate of official reports of child maltreatment, ascertained from records of the Missouri Department of Social Services at age 18 months. Child Maltreatment (number of cases of child abuse and neglect) as measured by official state administrative records

CONTACTS AND LOCATIONS:
Overall Officials: Mini Tandon, DO, Principal Investigator — Faculty
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Constantino JN. Child Maltreatment Prevention and the Scope of Child and Adolescent Psychiatry. Child Adolesc Psychiatr Clin N Am. 2016 Apr;25(2):157-65. doi: 10.1016/j.chc.2015.11.003. Epub 2016 Jan 11. PMID 26980121
- [Background] Jaffee SR. Child Maltreatment and Risk for Psychopathology in Childhood and Adulthood. Annu Rev Clin Psychol. 2017 May 8;13:525-551. doi: 10.1146/annurev-clinpsy-032816-045005. Epub 2017 Mar 30. PMID 28375720
- [Background] US DHHS, Children's Bureau (2017). Child Maltreatment 2015. Washington, DC: Author.U.S.
- [Background] Wu SS, Ma CX, Carter RL, Ariet M, Feaver EA, Resnick MB, Roth J. Risk factors for infant maltreatment: a population-based study. Child Abuse Negl. 2004 Dec;28(12):1253-64. doi: 10.1016/j.chiabu.2004.07.005. PMID 15607768
- [Background] Putnam-Hornstein, E., & Needell, B. (2011). Predictors of child protective service contact between birth and age five: An examination of California's 2002 birth cohort. Children and Youth Services Review, 33(8), 1337-1344.
- [Background] Gilbert R, Widom CS, Browne K, Fergusson D, Webb E, Janson S. Burden and consequences of child maltreatment in high-income countries. Lancet. 2009 Jan 3;373(9657):68-81. doi: 10.1016/S0140-6736(08)61706-7. Epub 2008 Dec 4. PMID 19056114
- [Background] Paulsell, D., Avellar, S., Sama Martin, E., & Del Grosso, P. Home Visiting Evidence of Effectiveness Review: Executive Summary. Office of Planning, Research and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services. 2011. Washington, DC.
- [Background] Jonson-Reid M, Kohl PL, Drake B. Child and adult outcomes of chronic child maltreatment. Pediatrics. 2012 May;129(5):839-45. doi: 10.1542/peds.2011-2529. Epub 2012 Apr 23. PMID 22529281
- [Derived] Tandon M, Jonson-Reid M, Constantino JN. Documenting Opportunity for Systematic Identification and Mitigation of Risk for Child Maltreatment. J Am Acad Child Adolesc Psychiatry. 2022 Nov;61(11):1313-1316. doi: 10.1016/j.jaac.2022.05.008. Epub 2022 Jun 8. PMID 35690303